CLINICAL TRIAL: NCT02822404
Title: Assessment of Cystatin C as a Tubular and Glomerular Marker of Nephrotoxicity in Pediatric Oncology
Brief Title: Description of the Cystatin C as an Early Nephrotoxic Bio-marker in Pediatric Oncology
Acronym: CysPed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11 308 03
Record Dates: First submitted 2016-02-03; First posted 2016-07-04 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Kidney Diseases
Keywords: kidney toxicity
MeSH Terms: conditions — Kidney Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Urinary and blood sample (Experimental): Urinary and blood samples for cystatin C dosage
  Interventions: Dietary Supplement: Urinary and blood sample for Cystatine dosage

INTERVENTIONS:
Dietary Supplement: Urinary and blood sample for Cystatine dosage — Urinary and blood cystatin C are sampled in patient with nephrotoxic risks before the treatment beginning, after the first course of chemotherapy, in the middle and at the end of the treatment. A follow up assessment is also required at 2 and 5 years. The cystatin C measurements are compared to traditional nephrology markers. Their sampling requires additional blood and urinary collection but involve minimal risks for patient.

SUMMARY:
Cisplatin and ifosfamide are commonly used drugs in chemotherapy. They are known to involve renal toxic threats in children given their immature kidney. This toxicity is increased especially after nephrectomy and/or concomitant radiotherapy. In pediatric oncology, the available evaluation methods of the renal function could be very restrictive to perform on children. In this study, the investigators intend to test the use of the cystatin C as an effective and reliable biological marker of renal toxicity in children treated with cisplatin and / or ifosfamide.

DETAILED DESCRIPTION:
Cisplatin and ifosfamide are commonly used drugs in chemotherapy. They are known to involve renal toxic threats in children given their immature kidney. This toxicity is increased especially after nephrectomy and/or concomitant radiotherapy. In pediatric oncology, the evaluation of the renal function is carried out according to the clinical trial protocols and to the center practices. To date, the standard methods (eg. creatinine clearance), as well as the available predictive formula (eg. Schwartz formula) are not well adapted to monitor children renal function. Indeed, the reliability of these methods depends on several parameters such as the diet and the muscle mass and could be very restrictive to perform on children. To circumvent these practical difficulties, the investigators intend to use the cystatin C as a biological marker of renal toxicity in children treated with cisplatin and / or ifosfamide. This cysteine protease has witnessed an upsurge of interest as an endogenous glomerular filtration rate marker and could be a good candidate to assess tubular toxicity when measured in urine.

This study aims to describe the kinetic of the appearance of the urinary cystatin C and explore its proprieties as an early and cost-effective marker for glomerular and tubular renal toxicity in children. In addition, this method could allow enhancing the calculation models routinely used for glomerular filtration rate.

ELIGIBILITY:
Inclusion Criteria:

* Children of 0 to18 years treated with cisplatin and / or ifosfamide in the hematology-oncology unit of Toulouse University Hospital of children regardless to the pathology they have been treated for
* Children with more than 4kg
* Written informed consent given by both parents or legal representative
* Patient covered by a social security agreement

Exclusion Criteria:

* Impossibility to monitor and follow up the patient until the foreseeable end of the treatment (geographic reasons, etc.)
* Contraindication to EDTA clearance performing

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2012-02-17 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-05-04 (Actual)

PRIMARY OUTCOMES:
Urinary cystatin C rate | 1 month
Urinary cystatin C rate | 6 months
  at T2a and T2b (at the middle of treatment). It can depend on pathology
Urinary cystatin C rate | 1 year
  at T3 (at the end of treatment)It can depend on pathology
Urinary cystatin C rate | 2 years
Urinary cystatin C rate | 5 years

SECONDARY OUTCOMES:
Sensibility, specificity and positive predictive value for urinary CysC | 5 years
  CysC is positive when it is detectable in urine, i.e when one or more reference biomarkers are positive
Predictive value for Glomerular Filtration Rate with blood rate of CysC (with Bouvet calculation method) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Marlène Pasquet, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lambert M, White-Koning M, Alonso M, Garnier A, Alphonsa G, Puiseux C, Munzer C, Berthier J, Malard L, Pasquet M, Chatelut E. Plasma cystatin C is a marker of renal glomerular injury in children treated with cisplatin or ifosfamide. Pediatr Blood Cancer. 2021 Jan;68(1):e28747. doi: 10.1002/pbc.28747. Epub 2020 Oct 15. PMID 33058496